CLINICAL TRIAL: NCT04518488
Title: Starting Recovery Pre-operatively: Feasibility of Implementing Individualized Prehabilitation for People Scheduled for Lower Limb Soft-tissue Sarcoma Surgery
Brief Title: Prehabilitation Soft-Tissue Sarcoma of Lower Limb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SARC-Prehab (2021-6796)
Record Dates: First submitted 2020-07-29; First posted 2020-08-19 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Soft Tissue Sarcoma
Keywords: prehabilitation; walking capacity; gait; quality of life
MeSH Terms: conditions — Sarcoma | interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Active Comparator): The prehabilitation group will receive a set of exercises designed to strengthen both limbs. The exercises will be taught and illustrated by a trained physiotherapist and are to be done daily during the period prior to surgery. The participant will be coached and supported for the exercise program, twice a week during the pre-operative period.
  Interventions: Other: Exercises
- Informational support group (control group) (Other): The focus for participants in the Informational Support Group will be on needs for information and psychosocial support during the pre-operative period. The intervention will be in the form of telephone or video calls by a trained health professional. These calls will be scheduled twice a week during the pre-operative period.
  Interventions: Other: Informational Support Group (Control group)

INTERVENTIONS:
Other: Exercises — Personalized and individualized exercises for lower limb soft-tissue sarcoma of each participant in this group.
  Arms: Prehabilitation group
Other: Informational Support Group (Control group) — The focus for participants in the Informational Support Group will be on needs for information and psychosocial support during the pre-operative period.
  Arms: Informational support group (control group)

SUMMARY:
This study is about preparing people with cancerous tumours, soft-tissue sarcoma (STS), in the leg to recover more quickly from surgery. Prehabilitation or "surgery school" is done before surgery while undergoing other cancer-related treatments. To test this idea, two groups will be formed. One group will have the prehabilitation program and the other group will have the same amount of attention from the research team who will visit them at the time of the radiotherapy sessions to provide support and any information they may need.The results of the study will indicate whether it is a good idea to conduct a bigger study that would involve many centres in Canada.

DETAILED DESCRIPTION:
This study is about preparing people with cancerous tumours, soft-tissue sarcoma (STS), in the leg to recover more quickly from surgery. Prehabilitation or "surgery school" is done before surgery while undergoing other cancer-related treatments. The tumour can be anywhere in the leg so exercises must be specially designed for each person. This process is novel and therefore has to be tested to see if it is practical and if it helps people recovery more quickly. To test this idea, two groups will be formed. One group will have the prehabilitation program and the other group will have the same amount of attention from the research team who will visit them at the time of the radiotherapy sessions to provide support and any information they may need. Assessments of how well participants can do basic activities of daily living will be assessed at study entry, just prior to surgery and then at 2, 6 and 12 weeks after surgery. Other measures of recovery will be distance covered while walking for six minutes, quality of the walking, and how quickly participants can walk outdoors for 1000 steps, and then 3000, 5000 and 9000. The investigators will ask participants which of these outcome measures they think best reflected their recovery and why. The investigators will also assess whether people were willing to enter the study and complete all the processes required. The results of the study will indicate whether it is a good idea to conduct a bigger study that would involve many centres in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Deep lower extremity Soft-tissue Sarcoma (buttock to foot)
* Histologically or cytologically-proven Soft-tissue Sarcoma (excluding superficial location) of the lower extremity.

Exclusion Criteria:

* Patients with metastatic disease (distant or nodal)
* both and upper and lower extremity involvement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Toronto Extremity Salvage Score | Assessments will be carried out prior to radiotherapy, pre-operatively, and at 2, 6 and 12 weeks post-operatively.
  self-report measure comprising 30 items (0-100; 0 worse, 100 better outcome)
Change in Six-Minute Walk Test | Assessments will be carried out prior to radiotherapy, pre-operatively, and at 2, 6 and 12 weeks post-operatively.
  Walking Capacity
Daily step count | 12 weeks
  will be obtained using the native accelerometer/gyroscope and pedometers available on both iphone (iOS) and android devices. For example, the android connection is through Google Fit
Change in Gait Quality (Angular velocity, cadence, heel strike) | Assessments will be carried out prior to radiotherapy, pre-operatively, and at 2, 6 and 12 weeks post-operatively.
  Obtained through device placed on the shoe of participants

SECONDARY OUTCOMES:
Change in Edmonton Symptom Assessment Scale | Assessments will be carried out prior to radiotherapy, pre-operatively, and at 2, 6 and 12 weeks post-operatively.
  7 symptoms including pain, fatigue, distress, and overall well-being (0-70; 0 better outcome; 70 worst outcome)
Change in health related quality of life | Assessments will be carried out prior to radiotherapy, pre-operatively, and at 2, 6 and 12 weeks post-operatively.
  Generic Quality of life (EQ-5D-5L)
Change in individualized health related quality of life | Assessments will be carried out prior to radiotherapy, pre-operatively, and at 2, 6 and 12 weeks post-operatively.
  Patient Generated Index

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mayo, PhD, Principal Investigator — Research Institute - MUHC

IPD SHARING:
Plan to Share IPD: Undecided